CLINICAL TRIAL: NCT00389051
Title: A Multicenter, Open Study to Assess the Tolerability, Pharmacokinetics and Antitumor Effect of Bendamustine Hydrochloride (SyB L-0501: 90 or 120 mg/m2/Day) Administered Intravenously for Two Days in Patients With Indolent Lymphoma
Brief Title: A Phase I Study of Bendamustine Hydrochloride in Patients With Indolent B-cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Katsuhisa Goto, SymBio Pharmaceuticals Limited
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006001
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2008-08

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Non-Hodgkin's Lymphoma; Malignant lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — Bendamustine Hydrochloride

INTERVENTIONS:
Drug: bendamustine hydrochloride — 1 cycle; 120 mg/m2/day,2 days concecutively, followed by 19days of oveservation period. (3 to 6 cycles)

SUMMARY:
The purpose of this study is to assess the tolerability, pharmacokinetics and antitumor effect of bendamustine hydrochloride (SyB L-0501) in patients with indolent B-cell Non-Hodgkin's Lymphoma.

DETAILED DESCRIPTION:
Indolent B-cell Non-hodgkin's lymphoma is treated mainly with radiation and chemotherapy using a combination of chemotherapies, such as purine-analogues and CHOP (cyclophosphamide, doxorubicin, vincristine and prednisolone). After the approval of an antibody therapy agent Rituximab®, it alone or combination with CHOP has been introduced. Bendamustine hydrochloride has a unique structure compared with the marketed agents, and has an innovative mechanism of action. Thus, it is expected that Bendamustine hydrochloride will provide new alternatives for patients with indolent B-cell Non-hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

Indolent B cell Non-Hodgkin's lymphoma patients with prior therapy who satisfy the conditions listed below. No restrictions regarding gender.

* Patients with histologically or cytologically confirmed indolent B cell Non-Hodgkin's lymphoma.
* Patients who had not received treatment (chemotherapy, antibody therapy and radiation/ radiotherapy) for more than 4 weeks following prior therapy and who are judged to carry no effect from the prior therapy.
* Patients aged from 20 to less than 75 years.
* Patients who had agreed in-patient during first course therapy.
* Patients from whom written consent to participate in this study has been obtained.

Exclusion Criteria:Patients who meet any of the following criteria will be excluded.

* Patients with apparent infections.
* Patients with serious complications (hepatic failure or renal failure).
* Patients with complication or history of serious heart failure (e.g. cardiac infarction, ischemic heart disease).
* Patients with serious digestive symptoms (nausea/ vomiting/ diarrhea).
* Patients who are known to be positive for HBV, HCV or HIC.
* Patients receiving other investigational drugs within 3 months before registration in the study.
* Patients with allogenic transplant.
* Women who are pregnant, of childbearing potential, or lactating.
* Patients who do not agree to contraception.
* Otherwise, patients who are judged by the investigator as being unsuitable for inclusion in the study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-10-31 (Actual); Primary Completion 2007-07-05 (Actual); Study Completion 2007-10-26 (Actual)

PRIMARY OUTCOMES:
Non-Hematological toxicity; > grade three(CTCAE v.3.0), during the treatment cycle (twenty one days)

SECONDARY OUTCOMES:
All adverse events or adverse reactions, during the treatment cycle (twenty one days)
Pharmacokinetics profile

CONTACTS AND LOCATIONS:
Overall Officials: Kensei Tobinai, MD, PhD, Study Chair — National Cancer Center Hospital
Locations (4):
- Japan (4):
  - Kanagawa
  - Kyoto
  - Nagoya
  - Tokyo

REFERENCES:
- [Derived] Ogura M, Uchida T, Taniwaki M, Ando K, Watanabe T, Kasai M, Matsumoto Y, Shimizu D, Ogawa Y, Ohmachi K, Yokoyama H, Tobinai K; Japanese Bendamustine Lymphoma Study Group. Phase I and pharmacokinetic study of bendamustine hydrochloride in relapsed or refractory indolent B-cell non-Hodgkin lymphoma and mantle cell lymphoma. Cancer Sci. 2010 Sep;101(9):2054-8. doi: 10.1111/j.1349-7006.2010.01633.x. PMID 20594195